CLINICAL TRIAL: NCT04301973
Title: Stools and Life Habits Collection in Heathy Volunteers/Subjects - to Provide Material for in Vitro Model Development
Acronym: PEPSIIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NU387
Record Dates: First submitted 2020-03-03; First posted 2020-03-10 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2020-12

CONDITIONS: Healthy Subjects
Keywords: Stool collection; Human samples collection; Healthy subject; Life habits questionnaires; Diet questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy people (Other)
  Interventions: Other: Stool collection

INTERVENTIONS:
Other: Stool collection — There is no intervention with a product in this study. The healthy subject has just to come 2 times in the clinical trial unit for clinical exam including urinary pregnancy test, fill life habits and diet questionnaires, and provide one stool sample for the 2nd visit, after 2 weeks of alimentary restrictions.

SUMMARY:
The purpose of this clinical study is to collect well characterized stools from healthy adult subjects, with completed life habits and alimentary questionnaires.

ELIGIBILITY:
Inclusion Criteria:

I1. Age between 18 and 69 years (limits included), I2. Body Mass Index (BMI) between 20 and 25 kg/m² (lower limit excluded and upper limit included), I3. Having regular Spontaneous Bowel Movements at the interview (a minimal of 7 SBMs per week is considered as regular);

I4. Ability to follow study procedures including at least:

* Stool collection, sampling, handling and storage throughout the duration of the study,
* Questionnaires and daily diet diary completion throughout the duration of the study,
* No substantial change in physical activity, diet regimen during the study period, I5. No prior medical consultation (primary or follow-up) for constipation or diarrhea, linked or not to infectious diseases, within the last 6 months; I6. Subject who accepts not to consume listed specific products including: yoghurts, fermented dairy products with probiotics and/or prebiotics, over-the-counter (OTC) medication containing probiotics and/or prebiotics, OTC medication such as herbal plants, psyllium, hormonal derivatives (e.g. melatonin, Dehydroepiandrosterone (DHEA) ...), food and nutritional supplements (e.g. vitamins and / or minerals such as Iron, Calcium and Magnesium) (called "prohibited products");

I7. For female subject: If woman of child bearing age, she must be using or complying with one of the following medically approved methods of contraception such as, but not exclusively:

1. Oral birth control pills at least 1 full monthly cycle prior to study;
2. Intra-uterine device (IUD);
3. Double barrier methods (such as condoms and spermicide); OR woman without contraception must be postmenopausal for at least 12 months prior to study entry or surgically sterile (i.e. hysterectomy, bilateral oophorectomy or bilateral tubal ligation).

I8. Good general health in the opinion of the investigator: no clinically significant and relevant abnormalities revealed by medical history or physical examination, I9. Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form, I10. Affiliated with a social security scheme, I11. Agree to be registered in the National biomedical research file for volunteers.

Exclusion Criteria:

E1. For female subject: pregnant woman or woman planning to become pregnant during the study or breast-feeding woman; E2. Ongoing - diagnosed gastrointestinal acute or chronic disease or complication (e.g; IBS, Crohn's disease, hemorrhoids, …);

E3. Previous (within one month), ongoing or planned therapy during the study with drugs altering bowel function:

* 5-HT3 receptor antagonists,
* Anticholinergic agents (tricyclic antidepressants, antiparkinsonian drugs, antipsychotics, antispasmodics, antihistamines),
* Anticonvulsants,
* Antihypertensives (calcium channel blockers, diuretics, centrally acting, antiarrhythmics, beta-adrenoreceptor antagonist),
* Bile acid sequestrants,
* Cation-containing agents (aluminum, bismuth, lithium),
* Chemotherapy agents (vinca alkaloids, alkylating agents),
* Laxatives or antidiarrheal drugs,
* Anti-Gastro- oesophageal reflux disease (GORD) medication
* Pain treatment/analgesics (opiates) except paracetamol or aspirin if occasional intake,
* Non-Steroidal Anti-Inflammatory Drugs (NSAID, including cortisone) if regular use
* Serotonin-Specific Reuptake Inhibitor (SSRI);
* Change of contraceptive method hormone replacement therapy for female subjects E4. Current or previous antibiotic, antifungal and antiparasitic treatment within 6 months; E5. Subject that have had any invasive diagnostic or therapeutic procedure(s) (except drawing blood), including dental surgery, with or without general or local anesthesia within the last 4 weeks or planned during the course of the study; E6. Subject with gastric or duodenal ulcer; E7. Shiftworker, subject going on holiday, subject planning to have its lifestyle habits modified (international travel, aircraft staff …) during study period; E8. Alcohol (consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women), drugs or medication abuse; E9. Known gluten intolerance, lactose intolerance and allergy to milk proteins; E10. Subject who stopped smoking, including the electronic cigarette, within 3 last months or intends to give up smoking during the study; E11. Subject who is following a special diet (e.g. slimming or vegetarian/vegan diets, medicated diet prescribed by a dietician or general practitioner such as a low cholesterol diet, low salt diet, low FODMAP, specific high-fiber diet, paleolithic or ketogenic diets…); E12. Subject enrolled in another clinical study in the last 30 days or in an exclusion period following participation in another clinical study; E13. Subject with severe life-threatening illness;

E14. Any significant systemic disease such as, but not limited to:

* Subjects who are currently suffering from an eating disorder such as anorexia or bulimia;
* Mechanical obstruction (colon cancer, external compression, strictures, postsurgical abnormalities, known megacolon, anal fissure);
* Metabolic conditions (diabetes mellitus, hypothyroidism, hypercalcemia, hypokalemia, hypomagnesia, uremia, heavy metal poisoning);
* Myopathies (amyloidosis, scleroderma);
* Neuropathies (Parkinson's disease, spinal cord injury or tumor, cerebrovascular disease, multiple sclerosis);
* History of asthma, hay fever, or other allergies;
* Other conditions (depression, degenerative joint disease, autonomic neuropathy, cognitive impairment, immobility, cardiac and cardiovascular diseases).

E15. Vulnerable subject defined as individual whose willingness to volunteer in the clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. (Examples are members of a group with a hierarchical structure linked to the Investigator or to the Sponsor, such as medical, pharmacy, dental and nursing students, subordinate hospital and laboratory personnel, employees of the Investigator or of the Sponsor, members of the armed forces, and persons kept in detention); E16. Having received, during the last 12 months, indemnities for clinical study higher or equal to 4500 Euros; E17. Subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject; E18. Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision; E19. Presenting a psychological or linguistic incapability to sign the informed consent; E20. Impossible to contact in case of emergency.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Characterized the consistency of stool collected from 4-days diet diary questionnaire after 14 days of dietary restrictions | After 14 days
Characterized the consistency of stool collected from the Intestinal Gas Questionnaire (IGQ) after 14 days of dietary restrictions | After 14 days
Characterized the consistency of stool collected from the Bristol Stool Scale (BSS) after 14 days of dietary restrictions | After 14 days

SECONDARY OUTCOMES:
Description of the dietary habits from the Food Frequency Questionnaire at Baseline | Baseline
Description of the life style habits from the International Physical Activity Questionnaire Short Form, at Baseline and after 14 days of dietary restrictions | Baseline and after 14 days
Description of the smoking habits from the tobacco questionnaire at Baseline | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Saint-Herblain, France